CLINICAL TRIAL: NCT00930969
Title: ST Segment Detection Study
Acronym: ST Detect
Status: Terminated | Type: Observational
Why Stopped: Low observed spontaneous coronary event rate among enrolled subjects
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: ST Detect
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Results first posted 2012-04-20 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac Ischemia; ST segment elevated Myocardial Infarction (STEMI); Non-ST Segment elevated Myocardial Infarction (NSTEMI); Implantable Cardioverter Defibrillator (ICD); Cardiac Electrogram (EGM); Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ICD — Subjects implanted with an ICD.

SUMMARY:
The purpose of ST Detect study is to evaluate whether naturally occurring spontaneous coronary events and exercise induced cardiac ischemia, give rise to detectable changes on intracardiac electrogram (EGM) signals in patients that are indicated for an Implantable Cardioverter Defibrillator (ICD) who have coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated for an ICD implantation
* AND subject must meet ONE of the following:

  * Prior acute coronary event
  * Previously underwent Percutaneous Coronary Intervention (PCI) or stent procedure
  * Multivessel disease
  * Positive stress test completed with evidence of ischemic heart disease, as determined by physician, and no subsequent successful revascularization

Exclusion Criteria:

* Subject is currently dependent on ventricular pacing
* Subject has Left Bundle Brunch Block (LBBB) and/or wide QRS
* Subject has chronic Atrial Fibrillation (AF)
* Subject has dementia
* Subject is indicated for a single chamber device
* Subject requires a right sided or abdominal ICD implant
* Subject is pregnant or in fertile age without secure birth control
* Subject has New York Heart Association (NYHA) class IV or refractory heart failure
* Subject is not expected to survive greater than 12 months
* Subject is participating in other confounding research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects coming into the hospital or the emergency room needing a defibrillator device having had coronary artery disease as outlined in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2008-04; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Crossley, MD, Principal Investigator — St. Thomas Research Institute and University of Tennessee College of Medicine Nashville, TN; Timothy Henry, MD, Principal Investigator — Minneapolis Heart Institute Foundation Minneapolis, MN
Locations (25):
- United States (17):
  - Anchorage, Alaska
  - Brandon, Florida
  - Orlando, Florida
  - Davenport, Iowa
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Mineola, New York
  - Stony Brook, New York
  - Gastonia, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Nashville, Tennessee
  - Austin, Texas
  - Burlington, Vermont
  - Richmond, Virginia
  - Morgantown, West Virginia
- Linz, Austria
- Liège, Belgium
- Copenhagen, Denmark
- Germany (3):
  - Berlin
  - Heidelberg
  - Nuremberg
- Zwolle, Netherlands
- Kristiansand, Norway

RESULTS

PARTICIPANT FLOW:
Groups:
- ICD Indicated: Subjects indicated for ICD therapy and at risk for recurrent myocardial infarction.
Period: Overall Study
Arm/Group | ICD Indicated
Started | 175
Completed | 137
Not Completed | 38
Not completed — Death | 5
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 13
Not completed — Withdrawal by Subject | 19

BASELINE CHARACTERISTICS:
Arm/Group | ICD Indicated
Number analyzed (Participants) | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 118
  >=65 years | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 147
Region of Enrollment [Number; unit: participants]
  United States | 134
  Denmark | 13
  Austria | 10
  Norway | 3
  Netherlands | 11
  Germany | 3
  Belgium | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ST Segment Changes During Myocardial Infarction
Description: The primary objective of the study was to observe if there are any detectable ST segment changes on an electrogram (EGM) signal from an implanted cardiac defibrillator (ICD) during myocardial infarctions among study participants.
Time Frame: Implant to 2 years
Population: During the study, none of the subjects presented with a ST Elevation Myocardial Infarction (STEMI). Therefore, there was not the opportunity to measure the hearts electrical activity during one of these events.
Arm/Group | ICD Indicated
Number analyzed (Participants) | 0

2. Secondary Outcome: Occurrence of Spontaneous Coronary Event
Description: During the study, spontaneous coronary ischemic events were categorized as STEMI, Non-ST elevated myocardial infarction (NSTEMI), or Unstable Angina. This objective was to provide estimates of rates per patient year for the study population. Rates are presented as: Average number of events per patient year (95% Confidence Interval)
Time Frame: Implant to 2 years
Population: There were 175 subjects that consented to participate in the study, and two subjects were not implanted with an ICD by the time the study was terminated. Therefore data collected by the implanted ICD in the remaining 173 subjects was analyzed.
Measure: Number (95% Confidence Interval); unit: Events per patient year
Arm/Group | ICD Indicated
Number analyzed (Participants) | 173
Events per patient year
  STEMI | 0 [0 to 2.1]
  NSTEMI | 2.9 [1.2 to 6.9]
  Unstable Angina | 5.1 [2.7 to 9.9]

3. Secondary Outcome: ST Segment Changes Measured by an ICD in Subjects Who Test Positive for Ischemia During an Exercise Stress Test
Description: Patients underwent an exercise stress test at their one month study visit. This objective was to summarize the magnitude of the hearts electrical activity signal measured by the implanted ICD during a positive exercise stress test for ischemia.
Time Frame: One-month follow-up visit
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | ICD Indicated
Number analyzed (Participants) | 18
millivolts | 1.23 (0.91)

4. Secondary Outcome: Number of Years of Stored Data in a Database of the Hearts Electrical Activity in This Specific Patient Population to be Used for Future Research.
Description: The device in this study included an additional capacity to collect and store information about the hearts electrical activity specific to ischemic heart disease. This additional capacity of the device is not currently available in market release ICDs. There is no measure to this objective, other than reporting the number of follow-up years of data accrued, which can be used by Medtronic for additional research.
Time Frame: Implant to 2 years
Population: There were 175 subjects that consented to participate in the study, and two subjects were not implanted with an ICD by the time the study was terminated. Therefore the number of years of stored device data to utilize for future research as collected by the implanted ICD in the remaining 173 subjects was analyzed.
Measure: Number; unit: Years
Arm/Group | ICD Indicated
Number analyzed (Participants) | 173
Years | 164.1

5. Secondary Outcome: Participants That Consented to Wear a Holter Monitor for a Period of 24 Hours to Collect Heart Sounds Data.
Description: When study subjects completed their six-month follow-up visit, they were asked if they would consent to wear a Holter monitor for a period of 24 hours to collect Heart Sounds data. The study subject would have to return to the center the following day to return the Holter monitor and have their ICD EGM vectors reprogrammed.
Time Frame: Six-month follow-up visit
Population: A subset of participants opting to wear a Holter monitor for 24 hours to collect Heart Sounds data, and then returning the following day for device reprogramming.
Measure: Number; unit: Participants
Arm/Group | ICD Indicated
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Baseline through 2 years.
Arm/Group | ICD Indicated
Serious Adverse Events (participants affected / at risk) | 86/175
Other Adverse Events (participants affected / at risk) | 20/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICD Indicated (N=175)
Angina pectoris (General disorders) | 11 (12)
Cardiac failure (General disorders) | 4 (12)
Cardiac failure acute (General disorders) | 5 (11)
Pneumonia (General disorders) | 5 (7)
Unstable angina (General disorders) | 9 (9)
Lead dislodgement (General disorders) | 5 (5)
NSTEMI (General disorders) | 4 (5)
Ventricular tachycardia (General disorders) | 4 (5)
Anaemia (General disorders) | 4 (4)
Chest pain (General disorders) | 5 (5)
Dyspnoea (General disorders) | 3 (4)
Chronic obstructive pulmonary disease (General disorders) | 3 (3)
Gastrointestinal haemorrhage (General disorders) | 3 (3)
Inappropriate device therapy (General disorders) | 2 (3)
Urinary tract infection (General disorders) | 3 (3)
Atrial fibrillation (General disorders) | 3 (3)
Atrial flutter (General disorders) | 2 (2)
Bleeding (General disorders) | 2 (2)
Cerebrovascular accident (General disorders) | 2 (2)
Cholecystitis acute (General disorders) | 2 (2)
Deep vein thrombosis (General disorders) | 4 (4)
Gastroenteritis (General disorders) | 2 (2)
Hypotension (General disorders) | 2 (3)
Implant site infection (General disorders) | 2 (2)
Intermittent claudication (General disorders) | 2 (2)
Ischaemic cardiomyopathy (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Pulmonary embolus (General disorders) | 2 (2)
Seizure (General disorders) | 1 (2)
Syncope (General disorders) | 2 (2)
Acute renal insufficiency (General disorders) | 1 (1)
Atelectasis (General disorders) | 1 (1)
Abdominal hernia (General disorders) | 1 (1)
Abscess (General disorders) | 1 (1)
Acute coronary syndrome (General disorders) | 1 (1)
Adenocarcinoma (General disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Ankle fracture (General disorders) | 1 (1)
Atrial tachycardia (General disorders) | 1 (1)
Bronchitis bacterial (General disorders) | 1 (1)
COPD Exacerbation (General disorders) | 1 (1)
Cardio-respiratory arrest (General disorders) | 1 (1)
Carotid artery stenosis (General disorders) | 1 (1)
Cellulitis (General disorders) | 1 (1)
Clostridium difficile sepsis (General disorders) | 1 (1)
Colitis ischaemic (General disorders) | 1 (1)
Colon cancer (General disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Diverticular perforation (General disorders) | 1 (1)
Diverticulum (General disorders) | 1 (1)
Dressler's syndrome (General disorders) | 1 (1)
Endocarditis (General disorders) | 1 (1)
Faecaloma (General disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gastritis (General disorders) | 1 (1)
Gout (General disorders) | 1 (1)
Hypotension (General disorders) | 1 (1)
Haematuria (General disorders) | 1 (1)
Haemoptysis (General disorders) | 1 (1)
Hepatitis C (General disorders) | 1 (1)
Hypersensitivity (General disorders) | 1 (1)
Hypertension (General disorders) | 1 (1)
Implant site hematoma (General disorders) | 1 (1)
Incision site hematoma (General disorders) | 1 (1)
Incisional hernia (General disorders) | 1 (1)
Infected hydrocele (General disorders) | 1 (1)
Infected sebaceous cyst (General disorders) | 1 (1)
Lower extremity edema (General disorders) | 1 (1)
Lymph node abscess (General disorders) | 1 (1)
Mental status changes (General disorders) | 1 (1)
Musculoskeletal pain (General disorders) | 1 (1)
Nasal septum deviation (General disorders) | 1 (1)
Neuralgia (General disorders) | 1 (1)
Obesity (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Oesophageal carcinoma (General disorders) | 1 (1)
Orthostatic hypotension (General disorders) | 1 (1)
Pneumothorax (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (General disorders) | 1 (1)
Pancreatitis (General disorders) | 1 (1)
Phimosis (General disorders) | 1 (1)
Post-traumatic headache (General disorders) | 1 (1)
Presyncope (General disorders) | 1 (1)
Radiculopathy (General disorders) | 1 (1)
Rectal cancer (General disorders) | 1 (1)
Renal artery stenosis (General disorders) | 1 (1)
Renal failure acute (General disorders) | 1 (1)
Renal mass (General disorders) | 1 (1)
Respiratory failure (General disorders) | 1 (1)
Respiratory tract infection (General disorders) | 1 (1)
Sepsis (General disorders) | 1 (1)
Sepsis MRSA (General disorders) | 1 (1)
Septic shock (General disorders) | 1 (1)
Skin laceration (General disorders) | 1 (1)
Spinal osteoarthritis (General disorders) | 1 (1)
Staphylococcal bacteraemia (General disorders) | 1 (1)
Stomach mass (General disorders) | 1 (1)
Thyroglossal cyst (General disorders) | 1 (1)
Traumatic fracture (General disorders) | 1 (1)
Urosepsis (General disorders) | 1 (1)
Ventricular fibrillation (General disorders) | 1 (1)
Wound haemorrhage (General disorders) | 1 (1)
Angina Unstable (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICD Indicated (N=175)
Atrial fibrillation (General disorders) | 8 (8)
Angina pectoris (General disorders) | 6 (7)
Dyspnea (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigational Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication.